CLINICAL TRIAL: NCT05208684
Title: Prolactin Release Through Breast Stimulation in Non-lactating Women - Who Does Respond?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRL Pilot
Record Dates: First submitted 2021-12-08; First posted 2022-01-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Prolactin; Breast Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast stimulation (Experimental): A 30-minute stimulation with moderate intensity by an electric milk pump (Elvie Pump) will be performed.
  Interventions: Other: Breast stimulation

INTERVENTIONS:
Other: Breast stimulation — Breast stimulation by the Elvie Pump to trigger prolactin release.

SUMMARY:
Prolactin is a multifunctional hormone which acts in different cell types rather than just modulating reproduction and lactation. One additional point is its action on glucose metabolism which is described especially in rodents. Prolactin affects proliferation, survival and insulin production of pancreatic beta cells in animal models. But also in human studies prolactin is linked to insulin action. Low systemic levels of prolactin are associated with increased prevalence of diabetes and while higher levels are associated with higher insulin sensitivity.

Acute metabolic effects of prolactin in young, healthy and non-lactating women should be accessed. Therefore, the induction of a transient increase of circulating prolactin levels is necessary to study the acute effects of this hormone on metabolic processes. This can most likely be achieved in non-pregnant and non-lactating women without pharmacological intervention.

As the main stimulus of prolactin release from the pituitary gland is the mechanical stimulation of the breast / nipple, like a suckling baby, stimulation by a breast pump might trigger prolactin release.

Due to other studies in this field, only a minority of women respond to breast stimulation with an increase in prolactin levels. Therefore, this pilot study will assess if an electric milk pump can stimulate prolactin release in non-lactating women. The second aim of the study is to identify factors which determine response and non-response to breast stimulation.

Prolactin will be measured in blood serum. The primary objective of this study is to identify women in whom a 30-minute breast stimulation causes a marked prolactin release. Response is defined as an increase at least twice the baseline value.

Second outcomes are the quantification and duration of prolactin increase as well as to detect differences in responders and non-responders. Therefore, demographic data as well as anthropometric data will also be assessed. A 10-minute electrocardiography and non-invasive measurement of resting energy expenditure by indirect calorimetry will also be performed. History of menstrual cycle, intake of contraceptive, parity and lactation experience will be recorded. Physical activity level and feeling of hunger will be assessed by questionnaires.

Feeling of hunger, resting energy expenditure, blood pressure, heart rate and body temperature will be assessed repeatedly to register differences before and after stimulation. Blood and urine samples will be assessed for safety.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged between 18 and 45 years
* premenopausal (women, who had menses at any time in the preceding 24 consecutive months)
* BMI < 25 kg/m²
* Ability to understand and voluntarily sign an informed consent document prior to any study related procedures

Exclusion Criteria:

* Type 1 or Type 2 diabetes
* Intake of medication which may affect prolactin levels (e.g. Metoclopramide, Methyldopa, opiates, cimetidine), except birth control pill/hormonal contraception known hyperprolactinemia or hyperthyroidism
* any other serious illness that might impact the results as judged by the investigator (e.g. malignant disease, coronary heart disease)
* Pregnant / breastfeeding women (weaning at least 6 month ago)
* plastic breast surgery (with detachment of milk ducts)
* allergy to BPA-free plastic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prolactin release - yes/no | Sample collection will be from 0 to 90 minutes
  The primary objective of this study is to identify women in whom breast stimulation causes a marked prolactin release. Response is defined as an increase at least twice the baseline blood value.

SECONDARY OUTCOMES:
Prolactin levels | Sample collection will be from 0 to 90 minutes
  Quantification, duration and trajectory of prolactin increase will be assessed by measuring prolactin levels in blood
Differences in subjects age | 1 minute
  Differences between responders and non-responders will be assessed: differences in age by recording birth date
Differences in subjects BMI | 4 minutes
  Differences between responders and non-responders will be assessed: differences in Body Mass Index by measuring height and weight of subjects and calculate the BMI
Differences in subjects body fat content | 3 minutes
  Differences between responders and non-responders will be assessed: differences in body fat content by bioelectrical impedance analysis
Differences in subjects menstrual cycle phase | 2 minutes
  Differences between responders and non-responders will be assessed: differences in phase of menstrual cycle by recording the menstrual history
Differences in subjects intake of hormonal contraception | 2 minutes
  Differences between responders and non-responders will be assessed: differences in intake of hormonal contraception recording intake of medication
Differences in subjects parity | 2 minutes
  Differences between responders and non-responders will be assessed: differences in parity by recording family history
Differences in subjects history of lactation | 2 minutes
  Differences between responders and non-responders will be assessed: differences in history of lactation experience by recording history of lactation
Differences in subjects heart rate variability parameters: time domain (beats per minute) | 10 minutes
  Differences between responders and non-responders and within subjects will be assessed: differences in the time domain by two 10-minute 3 lead ECG measurements before and after stimulation
Differences in subjects heart rate variability parameters: Root Mean Square of successive RR interval differences (RMSSD) | 10 minutes
  Differences between responders and non-responders and within subjects will be assessed: differences in RMSSD by two 10-minute 3 lead ECG measurements before and after stimulation
Differences in subjects heart rate variability parameters: Standard deviation of RR-intervals (SDNN) | 10 minutes
  Differences between responders and non-responders and within subjects will be assessed: differences SDNN by two 10-minute 3 lead ECG measurements before and after stimulation
Differences in subjects heart rate variability parameters: frequency domain parameters | 10 minutes
  Differences between responders and non-responders and within subjects will be assessed: differences in low (LF) and high (HF) frequency power by two 10-minute 3 lead ECG measurements before and after stimulation
Differences in subjects heart rate variability parameters: Low to high frequency power ratio | 20 minutes
  Differences between responders and non-responders and within subjects will be assessed: differences in LF/HF - Ratio by two 10-minute 3 lead ECG measurements before and after stimulation
Differences in subjects physical activity level | 10 minutes
  Differences between responders and non-responders will be assessed: differences physical activity level by questionnaire including the baecke index
Differences in subjects stress reaction | Sample collection will be from 0 to 90 minutes
  Differences between responders and non-responders will be assessed: differences in stress, measured by cortisol levels in blood
Changes in feelings of hunger through stimulation | 10 minutes
  Register change of feeling of hunger before and after stimulation by 15 questions on a five-point Likert scale survey about food cravings (FCQ-S)
Changes in resting energy expenditure through stimulation | 30 minutes (each 15 minutes)
  Register change of resting energy expenditure before and after stimulation by indirect calorimetry
Changes in blood pressure through stimulation | 4 minutes
  Register changes in blood pressure before and after stimulation using an automatic instrument with a digital readout
Changes in heart rate through stimulation | 4 minutes
  Register changes in heart rate before and after stimulation using an automatic instrument with a digital readout
Changes in body temperature through stimulation | 1 minute
  Register changes of body temperature before and after stimulation by an ear thermometer
Changes of Hypothalamic-Pituitary-Adrenal axis activity | 90 minutes
  Changes in Corticotropin levels are assessed by measurement in blood
Changes of Hypothalamic-Pituitary-Somatotropic axis activity | 90 minutes
  Changes in Somatotropin and insulin-like growth factor 1 levels are assessed by measurement in blood
Changes of Hypothalamic-Pituitary-Prolactin axis activity | 90 minutes
  Changes in Prolactin levels are assessed by measurement in blood
Changes of Hypothalamic-Pituitary-Thyroid axis activity | 90 minutes
  Changes in levels of Thyroid-stimulating hormone, Triiodthyronine and Thyroxine are assessed by measurement in blood
Changes of Hypothalamic-Pituitary-Gonadal axis activity | 90 minutes
  Changes in levels of Follicle stimulating hormone, Luteinizing hormone, estradiol and progesterone are assessed by measurement in blood

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Otfried-Mueller Str. 10, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.